CLINICAL TRIAL: NCT01002508
Title: Safety and Efficacy of Vaccination Against Influenza in Patients With Scleroderma
Brief Title: Influenza Vaccination in Patients With Scleroderma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Ira Litinsky, Tel Aviv Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0344-09
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-08

CONDITIONS: Influenza Vaccine in Scleroderma
Keywords: influenza vaccine scleroderma immunogenicity safety
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Influenza vaccine — One dose of influenza vaccine

SUMMARY:
The safety and efficacy of vaccination against influenza in patients with scleroderma is not clear. The objective of this study is to assess its safety and efficacy in 50 patients with scleroderma in comparison with 30 controls

DETAILED DESCRIPTION:
Fifty patients with scleroderma and 30 healthy , aged matched controls will participate in the study.

After signing informed consent, all subjects will be vaccinated with the inactivated split virion vaccine which recommended by the WHO this fall.

Patients will be evaluated at weel 0 and 6 weeks later. Clinical evaluation will be based on the modified Rodnan score, number of digital ischemic ulcers, presence of gastrointestinal and respiratory symptoms, number of swollen and tender joints, visual global evaluation of the physician , ESR and CRP Blood with be collected on the day of vaccination and 6 weeks later.

The immunogenicity of the vaccine will be tested by Haemagglutination inhibition (HI) test.

Influenza virus has two important surface glycoproteins: the haemagglutinin (HA) and the neuraminidase (NA). Antigenic classification and subtyping of influenza viruses is based on these two glycoproteins. HA plays a key role in virus cell entry by binding to cell surface receptors, which are found also on red blood cells of certain species. Binding to red cells results in haemagglutination, which can be observed as a carpet of agglutinated red cells at the bottom of a tube or microtitre well. In the HI test, antibody directed against the viral haemagglutinins block the virus from binding to the blood cells and thus inhibits the haemagglutination reaction.

The pre- and post immunization HI antibodies were tested at the Central Virology Laboratory of the Israeli Ministry of Health using the HI test according to a standard WHO procedure 16. Sera were separated, code labeled, and stored at -20°C until tested. Sera were treated with receptor destroying enzyme cholera filtrate to remove non-specific inhibitors, and with Turkey red blood cells to remove non-specific agglutinins. The treated sera were tested by HI test against the three antigens included in the vaccine: A/California (CAL), A/Wisconsin and B/Malaysia. The working dilution (test dose) of each antigen contained four haemagglutinin units in 25 µl of antigen. Test doses were diluted in phosphate buffered saline (PBS) and added to serial dilution of antiserum. The haemagglutinin inhibition titer was determined as the highest dilution of serum that completely inhibits haemagglutination of red blood cells.

The titer of an antiserum not showing any inhibition will be recorded as <10. Humoral response will be defined as either a fourfold or more rise in titer, or a rise from a non-protective baseline level of <1/40 to 1/40 in HI antibodies four weeks after vaccination 17,18. Geometric mean titers of antibody will be calculated to assess the immunity of the whole group.

Primary Endpoint of the study : the proportion of patients who achieve a titer of antibodies above 1/40, against each of the antigens included in the vaccine Secondary Endpoint: Safety of the vaccine

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year old age
* Capable to sign a informed consent
* Suffering from scleroderma

Exclusion Criteria:

* Known allergy to influenza vaccine
* Allergy to eggs

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who achieve a titer of antibodies above 1/40 | 6 weeks

SECONDARY OUTCOMES:
Number of patients with an increased Rodnan Score | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Setti M, Fenoglio D, Ansaldi F, Filaci G, Bacilieri S, Sticchi L, Ferrera A, Indiveri F, Ghio M. Flu vaccination with a virosomal vaccine does not affect clinical course and immunological parameters in scleroderma patients. Vaccine. 2009 May 26;27(25-26):3367-72. doi: 10.1016/j.vaccine.2009.01.078. Epub 2009 Feb 5. PMID 19200840